CLINICAL TRIAL: NCT03994900
Title: A Monocentric Study Assessing the Efficacy of the Nitrosylated Hemoglobin as Biomarker for Detecting the Development of a Cardiovascular Complication During or After Surgery
Acronym: PICA
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Université Catholique de Louvain (Other)
Collaborators: SPINOVIT (Unknown)
Responsible Party: Principal Investigator, Jean-Luc Balligand, Professor MD, Université Catholique de Louvain
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: PICA V2.2
Record Dates: First submitted 2019-06-19; First posted 2019-06-21 (Actual); Last update posted 2022-11-21 (Actual); Status verified 2022-11

CONDITIONS: Cardiovascular Complications
Keywords: cardiovascular nitric oxide erythrocyte
MeSH Terms: interventions — Blood Specimen Collection

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Blood sampling for HbNO assessment (Experimental)
  Interventions: Diagnostic Test: Blood sampling for HbNO assessment

INTERVENTIONS:
Diagnostic Test: Blood sampling for HbNO assessment — Blood sampling

SUMMARY:
Cardiovascular diseases are the first mortality cause in Occidental countries. Surgery and anesthesia can provoke hemodynamic instability and stimulation of the sympathetic nervous system as well as bleeding or thrombosis. These factors as top of some post-operative factors such as tissular hypoxemia, can result in cardiovascular complications. Developing a tool to predict post-operative cardiovascular complication could influence peri-operative measures by stratifying the population at risk. UCLouvain has developed a patented technique using a paramagnetic electronic resonance spectrometry (EPR) able to quantify a paramagnetic component, nitrosylated hemoglobin (HbNO) of the erythrocytes drawn from venous blood. This HbNO has been correlated to the traditional cardiac risk factors. In this study, we will assess the HbNO of patients prior to surgery and will correlate it with cardiovascualr and non cardiovascular complications in order to evaluate the predictive aspect of our biomarker.

DETAILED DESCRIPTION:
Cardiovascular diseases are the first mortality cause in Occidental countries. They would be the cause of 31% of the overall mortality in those countries.

Some risk factors are strongly related to the apparition of a cardiovascular disease, including smoking, high cholesterol levels, hypertension, diabetes, age, high BMI or familial early cardiovascular disease and/or hypercholesterolemia.

Multiple studies have already shown that major non-cardiac surgery can lead to cardiovascular complications in 3% of the patients regardless of their cardiovascular risk profile and major adverse cardiovascular events are a significant source of post-operative morbidity in approximately 11% among those patient3,4,6,7. Complications can also lead to a prolongated hospitalization for patients undergoing major non-cardiac surgery8,9.The peri- and post-operative cardiovascular complications depend on patient-related risk factors.

Surgery and anesthesia can provoke hemodynamic instability and stimulation of the sympathetic nervous system. Surgery and the ensuing inflammation can also induce bleeding and or thrombosis. These factors as top of some post-operative factors such as tissular hypoxemia, can result in cardiovascular complications.

An assessment of the medical cardiac history of the patients is performed before any surgery3. Developing a tool to predict post-operative cardiovascular complication could influence peri-operative measures by stratifying the population at risk.

It is known that cardiovascular diseases are preceded by a dysfunction of the vascular endothelium leading to a loss of the antithrombogenic, anti-proliferative and vasorelaxant functions.

A key mediator of vascular homeostasis and endothelial integrity is the nitric oxide (NO) produced by the endothelial NO synthetase (eNOS). UCLouvain has developed a patented technique using a paramagnetic electronic resonance spectrometry (EPR) able to quantify a paramagnetic component, nitrosylated hemoglobin (HbNO) of the erythrocytes drawn from venous blood. This HbNO has been correlated to the traditional cardiac risk factors.

Quantifying the HbNO could predict, prior to any major non-cardiac surgery, an eventual peri-operative cardiovascular complication. Preoperative HbNO would as such be a useful marker of cardiovascular complications. Necessary perioperative measures can therefore be taken in order to decrease this risk. This assessment would be associated to the preoperative anesthesia visit (EPI : évaluation péri-interventionnelle) form reporting previous cardiovascular events and risk factors.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 and 100 years
* Written informed consent
* For subjects unable to read and/or write, oral informed consent observed by an independent witness is acceptable if the subject has fully understood oral information given by the Investigator. The witness should sign the consent form on behalf of the subject.
* Forthcoming major surgery + one of the following:

At least one risk factor for cardiovascular disease:

SCORE > 1% and < 5% BMI > 30 Age > 55 years BP: >130 SBP and/or >85 DBP Diabetes type 1 or 2 Active smoker regardless of age Shorteness of breath after climbing 20 stairs Familial early CV disease (<50 years for men; <55 years for women) Familial hypercholesterolemia (segregation of hypercholesterolemic trait or proven genetic mutation at heterozygous or homozygous state)

* LEE score >2
* Thrombophilia: Factor V Leiden
* Flap surgery
* Surgery for liver or kidney graft
* Known cause (i.e. COPD) of respiratory dysfunction; patients under positive pressure (CPAP) treatment
* Sleep apnea syndrome
* Pregnant women at risk of pre-eclampsia: > 20 weeks of pregnancy and one of the following:

SBP > 160 mmHg DBP > 110 mmHg Rise of SBP > 30 mmHg compared to baseline value Rise of DBP > 10 mmHg compared to baseline value Proteinuria ≥ 30 mg/L

o Pre-operative creatinine > 130 µmol/L (> 1.5 mg/dL)

Exclusion Criteria:

* Patients undergoing a cardiovascular surgery
* Patients unable to give informed consent (people under legal guardianship)
* Patients placed in an institution by official or court order

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2500 (Estimated)
Dates: Start 2019-10-01 (Actual); Primary Completion 2023-06-30 (Estimated); Study Completion 2023-09-01 (Estimated)

PRIMARY OUTCOMES:
Incidence of intra and postoperative cardiovascular complication or degradation within 12 months | 12 months
  Incidence of intra and postoperative cardiovascular complication or degradation within 12 months
the duration of hospitalization | 12 months
  the duration of hospitalization
the duration of residence in intensive care | 12 months
  the duration of residence in intensive care
the need for a follow-up by a cardiologist | 12 months
  the need for a follow-up by a cardiologist

SECONDARY OUTCOMES:
Incidence of a non-cardiovascular complication | 12 months
  Incidence of a non-cardiovascular complication
the LEE score at first visit | 12 months
  the LEE score at first visit

CONTACTS AND LOCATIONS:
Locations (1):
- Cliniques Universitaires St Luc, Brussels, Belgium

IPD SHARING:
Plan to Share IPD: No